CLINICAL TRIAL: NCT00386113
Title: A Phase II, Open, Controlled Study to Evaluate the Reactogenicity and the Immunogenicity of GlaxoSmithKline Biologicals' Adjuvanted Influenza Vaccine in Elderly Adults Previously Vaccinated With Either Fluarix™ or the Adjuvanted Vaccine.
Brief Title: Study to Evaluate Reactogenicity and Immunogenicity of Revaccination With Adjuvanted Influenza Vaccine in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107973
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Influenza
Keywords: Influenza; improved vaccine; elderly
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

INTERVENTIONS:
Biological: Fluarix and adjuvanted influenza vaccine

SUMMARY:
Since influenza vaccines are normally administered every year because of the frequent change in their antigenic composition, the safety and immunogenicity profile of adjuvanted influenza vaccine need to be re-evaluated after repeated vaccine administration. In this study, subjects previously vaccinated with Fluarix or the influenza adjuvanted vaccine, will receive a booster dose with the 2006-2007 season's formulations of either Fluarix or the adjuvanted vaccine.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be healthy elderly >/= 67 years and previously vaccinated with Fluarix or the adjuvanted vaccine.

Exclusion Criteria:

* Subjects will be excluded if they take/have taken chronically high doses of immunosuppressants or other immunemodifying drugs within six months before vaccination, or immunoglobulins or blood products within three months before vaccination, or any investigational product within 30 days before vaccination, have a history of influenza infection since previous vaccination, or if subjects have acute or chronic clinically significant disease or an immunosuppressive/deficient condition, or have contra-indications to influenza vaccination

Min Age: 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-10-16 (Actual); Primary Completion 2006-11-14 (Actual); Study Completion 2006-11-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and reactogenicity of repeated vaccination with adjuvanted influenza vaccine, during 21 days following administration of the vaccine.

SECONDARY OUTCOMES:
Evaluation of the humoral immune response & cell-mediated immune response 21 days after revaccination with candidate vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium